CLINICAL TRIAL: NCT00043576
Title: A Phase 2/3 Multicenter, Randomized, Double Blind Study of Docetaxel (Taxotere) Plus DN-101 or Placebo in Androgen Independent Prostate Cancer (AIPC)
Brief Title: ASCENT: Androgen Independent Prostate Cancer Study of Calcitriol Enhancing Taxotere
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novacea (Industry)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DN101-002; ASCENT Trial
Record Dates: First submitted 2002-08-09; First posted 2002-08-13 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2005-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Docetaxel

INTERVENTIONS:
Drug: calcitriol
Drug: docetaxel

SUMMARY:
The purposes of this study are to determine if DN-101 plus Taxotere lowers PSA levels, delays or limits disease progression and is safe with minimal side effects.

DETAILED DESCRIPTION:
DN-101 is an investigational drug that has not been approved by the U.S. Food and Drug Administration (FDA). It is a newly formulated pill that contains high amounts of calcitriol, a naturally occurring hormone and the biologically active form of vitamin D. Administration of DN-101 results in much higher blood levels of calcitriol than the body can produce from dietary vitamin D or vitamin D supplements. These higher levels of calcitriol are associated with anti-cancer effects in laboratory models of human cancer. Laboratory models also indicate that calcitriol has synergy with many commonly used chemotherapeutic agents used to treat cancer.

Calcitriol, at very low doses, is currently approved for use in patients with chronic kidney failure. DN-101 was specifically designed for cancer and contains 30 times the amount of calcitriol found in the calcitriol pill commercially available today. In order to take an amount of calcitriol equivalent to 1 DN-101 pill, cancer patients would need to swallow 30 pills of the approved, low dose formulation. DN-101 represents a breakthrough in the use of calcitriol in the clinic, because it contains high concentrations of calcitriol and makes it more feasible for patients to stay on regimen.

ELIGIBILITY:
* Three rising PSA measurements OR a new metastatic lesion
* Adequate liver and kidney function
* Ongoing hormonal therapy
* No hospitalization for angina, heart attack or congestive heart failure within the last 12 months
* No kidney stones in the last 5 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2002-08; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, MD, Study Chair — Oregon Health and Science University
Locations (62):
- United States (52):
  - Montgomery Cancer Center, Montgomery, Alabama
  - Arizona Cancer Center- Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center/Southern Arizona VA HCS, Tucson, Arizona
  - Arizona Cancer Center- Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences / Central AR VA, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - California Cancer Care, Greenbrae, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Prostate Oncology Specialist/Pacific Clinical Research, Marina del Rey, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Southern California Permanente Medical Group, San Diego, California
  - Sharp Healthcare, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Kaiser- Northern California, Vallejo, California
  - San Diego Cancer Center, Vista, California
  - Oncology Hematology Associates, Paudre Calley Cancer Ctr., Fort Collins, Colorado
  - University of Miami-Sylvester Comprehensive Cancer Center, Miami, Florida
  - Oncology Hematology Consultants, Sarasota, Florida
  - Georgia Urology, P.A., Atlanta, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Loyola University Medical, Maywood, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Urologic Associates- P.C., Davenport, Iowa
  - Oncology Hematology Care, Crestview Hills, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Associates in Oncology Hematology P.C., Rockville, Maryland
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Univ. of Nebraska Medical Center/VA Hospital, Omaha, Nebraska
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Union State Bank Cancer Center, Nyack, New York
  - Lincoln Medical & Mental Health Center, The Bronx, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - The Cleveland Clinic Foundation, Taussig Cancer Center, Cleveland, Ohio
  - Mid Ohio Oncology Hematology, Inc., Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - NW Kaiser Permanente Portland, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina
  - University Oncology/ Hematology Associates, Chattanooga, Tennessee
  - Boston Baskin Cancer Group, Memphis, Tennessee
  - Professional Quality Research, Austin, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Cancer Care, Fort Worth, Texas
  - Urology Associates of North Texas, Fort Worth, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Tyler Cancer Center, Tyler, Texas
  - University of Washington Cancer Care, Seattle, Washington
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Cancer Center, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Toronto-Sunnybrook Regional Cancer Center, Toronto, Ontario
  - Princess Margaret Hospital, University Health Network, Toronto, Ontario
  - CHUM / Notre-Dame Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Quebec, Hotel-Dieu de Quebec, Québec, Quebec

REFERENCES:
- [Background] Beer TM, Munar M, Henner WD. A Phase I trial of pulse calcitriol in patients with refractory malignancies: pulse dosing permits substantial dose escalation. Cancer. 2001 Jun 15;91(12):2431-9. PMID 11413535
- [Background] Beer TM, Eilers KM, Garzotto M, Egorin MJ, Lowe BA, Henner WD. Weekly high-dose calcitriol and docetaxel in metastatic androgen-independent prostate cancer. J Clin Oncol. 2003 Jan 1;21(1):123-8. doi: 10.1200/jco.2003.05.117. PMID 12506180